CLINICAL TRIAL: NCT05368168
Title: Impact of Early Postoperative Treatment With Posterior Tibial Nerve Stimulation on the Incidence and Duration of Low Anterior Rectal Resection Syndrome
Acronym: LARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Innovacion en Cirugía Vigo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LARS
Record Dates: First submitted 2022-05-04; First posted 2022-05-10 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Rectal Disorders; Low Anterior Resection Syndrome; Low Anterior Resection
Keywords: Posterior tibial nerve stimulation (PTNS); Urgent PC; Transcutaneous neurostimulator
MeSH Terms: conditions — Rectal Diseases; Low Anterior Resection Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Assignment to one group or the other will be randomized by a simple 1:1 randomization method through the CRF automatically and after hospital discharge.
  Double-blind masking will be performed (patients will not know to which group they belong and the investigator will not know to which group each patient is assigned). The only person aware of the outcome of the randomization will be the functional tests nurse, who will apply the PTNS treatment.
  Patients in both groups will be appointed in the same way in the functional testing office, although patients in group 2 will not receive PTNS, the tibial nerve puncture will be applied, they will be stimulated until they perceive the corresponding current and then the neurostimulator will be turned off so that they do not receive the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Posterior tibial nerve stimulation (PTNS) (Experimental): Patients operated on at the Hospital Álvaro Cunqueiro for rectal neoplasia with anastomosis below 10 cm and who, after randomization, WILL BE treated with posterior tibial nerve stimulation.
  Interventions: Device: Posterior tibial nerve stimulation (PTNS)
- Group 2: Standard of care (No Intervention): Patients operated on at the Hospital Álvaro Cunqueiro for rectal neoplasia with anastomosis below 10 cm and who, after randomization,WILL NOT BE treated with posterior tibial nerve stimulation.

INTERVENTIONS:
Device: Posterior tibial nerve stimulation (PTNS) — Posterior tibial nerve neurostimulation in postoperative patients treated for rectal neoplasms for 6 weeks at a rate of 2 sessions per week (12 sessions).
  The sessions will be carried out by the nursing staff of the anorectal functional testing cabinet. The sessions will begin 3 weeks after hospital discharge for patients without lateral ileostomy and after ileostomy closure for patients with lateral ileostomy.
  Other Names: Transcutaneous neurostimulator (Urgent PC)
  Arms: Group 1: Posterior tibial nerve stimulation (PTNS)

SUMMARY:
The treatment of rectal cancer is currently based on surgical resection of the rectum with total excision of the mesorectum, associated with neoadjuvant radiochemotherapy.

Surgical resections with sphincter preservation are frequently (60% of cases) associated with problems related to intestinal and defecatory function, which together are called Anterior Resection Syndrome (ARS) with varying degrees of severity.

Among the different treatments the investigators find posterior tibial nerve stimulation, a simple and non-invasive technique, which is currently used.

The study aims to analyze whether postoperative posterior tibial nerve stimulation in patients undergoing low anterior resection of the rectum has an impact on the incidence and duration of low anterior resection syndrome (LARS) and therefore on the quality of life of patients undergoing this type of intervention.

Therefore, treatment with PNTS is currently established for the management of LARS symptoms. Given that a large percentage of patients operated on for rectal neoplasms will develop this syndrome, the investigators intend to apply this treatment before the onset of symptoms in patients at risk for LARS. It is also an intervention with a low rate of side effects, the benefit that the investigators can obtain from its preventive application is clearly superior to the risk of undergoing such treatment.

The investigators´ hypothesis is: Posterior tibial stimulation for 6 weeks post-operative of low anterior resection with anastomosis has a favorable impact by reducing the incidence and duration of ARS and improving the quality of life of patients undergoing anterior rectal resections for cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery (scheduled, non-urgent) who underwent anterior rectal resection or transit reconstruction with low anastomosis (below 10 cm from the anal margin) at the Hospital Álvaro Cunqueiro in Vigo after the start date of the study.
* Anastomotic tightness (absence of dehiscence).
* Patients older than 18 years old.
* Acceptance to participate in the study.

Exclusion Criteria:

* Inability to understand the study instructions and recommendations.
* Dementia or any type of mental disability.
* Palliative surgery.
* Patients with pacemakers.
* Anti-coagulated patients.
* Patients with trophic lesions on the skin of the ankles.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of PTNS (Posterior Tibial Nerve Stimulation) treatment on the incidence and duration of RAS symptoms in patients undergoing anterior rectal resection with sphincter-sparing surgery. | 12 months
  Variables:
  Age (years), Sex (F/M), Gestation (Y/N), Births (Y/N), Tumor location (cm from anus), Radiotherapy (Y/N), Radiotherapy regimen (short/long), Neoadjuvant chemotherapy (Y/N), Surgical approach (open, laparoscopic,transanal/converted), Distance between anus and anastomosis (cm), Type of anastomosis (colorectal, coloanal, mechanical, manual, term-terminal, term-lateral), Performance of derivative stoma (Y/N), Extent of mesorectal excision (total/partial), Postoperative dehiscence (Y/N), Postoperative abdominal collection(Y/N). Postoperative bleeding (Y/N), Clavien-dindo classification.
  Time from surgery to stoma closure (months), sphincter disruption (Y/N), Manometry (mmHg), neurostimulation parameters: stimulation intensity (mA), foot (right/left), stimulus (sensitive/motor/both). LARS score (0-42)
Impact of PTNS on the quality of life (EORTC-QLQ C30) | 12 months
  To evaluate the impact of PTNS on the quality of life of patients undergoing anterior rectal resection with sphincter-sparing surgery (as assessed by the EORTC-QLQ C30 quality of life questionnaire).
  The "European organization for reseach and treatment of cáncer quality life questionnaire core 30" (EORTC-QLQ C30) is a cancer-specific, multidimensional questionnaire comprising 30 items on five scales (physical, functional, emotional, cognitive, social), three items on symptoms (fatigue, nausea/vomiting, pain), six single-item items (constipation, diarrhea, hyporexia, insomnia, dyspnea,economic difficulties) and others on a global state of health.
  The score is between 1 and 100, where the higher the score, the greater the decrease in quality of life.

SECONDARY OUTCOMES:
LARS Scale | 12 months
  To evaluate continence and number of stools (assessed by the LARS scale) in patients undergoing anterior rectal resection.
  "Low Anterior Resection Score" LARS scale is a quantitative variable of anterior resection syndrome related to quality of life. The scale ranges from 0 to 42 points with the highest score being a worsening result and it is categorized into 3 groups: no LARS (0-20 points), minor LARS (21-29 points) and major LARS (30-42 points).
Impact of PTNS on the quality of life (EORTC-QLQ C29) | 12 months
  To evaluate sexual dysfunction in patients undergoing anterior rectal resection (assessed by the European Organization for Research and Treatment of Cancer-Quality of Life Questionnaires: EORTC-QLQ C29).
  The "European organization for reseach and treatment of cáncer quality life questionnaire core 29" (EORTC-QLQ C29) is a questionnaire specific to patients with rectal neoplasms. It comprises 19 questions common to all patients, four questions on female or male sexual dysfunction and seven questions for patients with or without stoma.
  The score is between 1 and 136, where the higher the score, the greater the decrease in quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Sánchez Santos, PhD, Study Director — Complejo Hospitalario Universitario de Vigo
Locations (1):
- Hospital Álvaro Cunqueiro, Vigo, Pontevedra, Spain